CLINICAL TRIAL: NCT03220932
Title: Assessment of Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy in First or Secondary Platinum-resistant Recurrent Ovarian Epithelial Cancer
Brief Title: Cytoreductive Surgery and HIPEC in First or Secondary Platinum-resistant Recurrent Ovarian Epithelial Cancer
Acronym: HIPOVA-01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL17_0342
Record Dates: First submitted 2017-05-11; First posted 2017-07-18 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Ovarian Epithelial Cancer
Keywords: Epithelial Ovarian Cancer - Platinum-resistant - Cytoreductive surgery - HIPEC - Quality of Life
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Hyperthermic Intraperitoneal Chemotherapy; Drug Therapy; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cytoreductive surgery combined with HIPEC (Experimental): All patients will start with three cycles of CT-BEV 15 mg/kg, and will then be randomly. Then one cycle of monochemotherapy without bevacizumab is administered and followed by an interval CRS and HIPEC with postoperative chemotherapy and bevacizumab (CT-BEV - 15 mg/kg once every 3 weeks) until disease progression
  Interventions: Procedure: Cytoreductive surgery combined with HIPEC
- Aurelia arm (Active Comparator): Chemotherapy and bevacizumab (CT-BEV) once every 3 weeks from enrollment until disease progression
  Interventions: Drug: Chemotherapy and bevacizumab (CT-BEV)

INTERVENTIONS:
Procedure: Cytoreductive surgery combined with HIPEC — Cytoreductive surgery combined with HIPEC (Cisplatin 70 mg/m2).
  Arms: Cytoreductive surgery combined with HIPEC
Drug: Chemotherapy and bevacizumab (CT-BEV) — Chemotherapy and bevacizumab (CT-BEV) 15 mg/kg once every 3 weeks from enrollment until disease progression (RECIST 1.1)
  Arms: Aurelia arm

SUMMARY:
With 4,600 new cases in France in 2012, ovarian cancer is the seventh most common cancer in women and the fourth cause of mortality by cancer. Despite a high response rate to initial treatment, most patients will relapse within 2 years. No standard treatment has yet been established for patients with recurrent ovarian cancer.

Most patients with such recurrences are currently treated with new combinations of systemic chemotherapy. A repeated laparotomy with complete cytoreduction is also an option that several authors have used to obtain median survival rates of more than 30 months.

Twenty five percent of patients experiencing relapse present with platinum-resistant recurrence, occurring less than 6 months after chemotherapy completion. Recently, Pujade et al. showed that adding bevacizumab to chemotherapy significantly improves progression-free survival (PFS) in this subgroup of patients with poor prognoses (16.6 months versus 13.3 months in women treated with chemotherapy alone). Three case control studies have compared systemic chemotherapy and CRS (Cytoreduction Surgery) alone versus CRS plus HIPEC in patients with recurrent disease. They showed significantly improved results with the addition of HIPEC. In the French registry that included 474 patients with recurrence and peritoneal carcinomatosis, the median PFS was 13.8 months for platinum-resistant patients and 13 months for platinum-sensitive patients. Our hypothesis is that surgery would reduce the tumor burden and consequently the number of platinum-resistant tumor clones and that HIPEC would control the microscopic residual disease by increasing the tumor cell cytotoxicity.

We assume that adding a locoregional treatment to an "Aurelia-like" systemic treatment would improve the PFS. We aim to assess the benefit of adding surgery and HIPEC to the treatment of first or second platinum-resistant recurrence compared to chemotherapy + bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed platinum-resistant Epithelial Ovarian Carcinoma (EOC)(clinical recurrence or persistence within 6 months of last treatment);
* White blood cells >3,500/mm3, neutrophils ≥1,500/mm3, platelets ≥100,000/mm3;
* Good renal function: serum creatinine values <1.5 mg/dl, creatinine clearance >60 ml/min;
* Performance Status ≤2, Karnofsky Index ≥70%;
* Serum bilirubin ≤1.5 x Upper limit of normal (UNL) 2 mg/dl;
* Prior ovarian surgery before starting study treatment;
* Covered by a Healthcare System, where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research;
* Signed written informed consent obtained prior to any study-specific screening procedures.

Exclusion Criteria:

* Platinum-refractory EOC (i.e progression under platinum containing chemotherapy);
* Any prior malignancy not considered in complete remission for at least 2 years;
* Pregnancy or breastfeeding;
* Untreated central nervous system disease or symptomatic central nervous system metastasis, history or evidence of thrombotic or hemorrhagic disorders within 6 months before first study treatment;
* Uncontrolled hypertension or active clinically significant cardiovascular disease;
* Females of childbearing age not using medically accepted contraceptive measures, as judged by the investigator;
* Contraindication to any drug contained in the chemotherapy regimen;
* Known contraindication to cisplatin
* Medical, geographical, sociological, psychological or legal conditions that would prevent the patient from completing the study or signing the informed consent;
* Any significant disease which, in the investigator's opinion, excludes the patient from the study;
* Under any administrative or legal supervision.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-11-30 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Change from baseline to 36 months
  Progression will be based on RECIST V1.1 criteria performed on thoraco-abdominopelvic tomodensitometry (TDM ) assessed every 3 months. There is a follow-up period of 36 months.

SECONDARY OUTCOMES:
Overall survival | From the randomization to the death or 36 months end of follow-up
  There is a follow-up period of 36 months.
Potential treatment-related mortality | During the first 60 postoperative days
  Reported only in the experimental arm (cytoreductive surgery + HIPEC)
Potential treatment-related morbidity | During the first 60 postoperative days
  Adverse events (AE) during the follow-up period: safety and tolerability will be assessed in terms of AEs, deaths, laboratory data, and vital signs. AEs will be described using MedDRA terms (version 18.0) and graded according to Common Terminology Criteria for Adverse Events (CTCAE version 5.0). These will be collected for all randomized patients.
Quality of life assessment | Baseline to 36 months end of follow-up
  Quality of Life will be assessed using the Functional Assessment of Cancer Therapy-Ovarian (FACT-O) for all randomized patients.

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - Centre Hospitalier Universitaire Jean Minjoz, Besançon
  - Centre Oscar Lambret, Lille
  - CHRU Claude Huriez, Lille
  - Centre Léon Bérard, Lyon
  - Institut du Cancer de Montpellier, Montpellier
  - Centre Hospitalier Universitaire L'Archet II, Nice
  - Hôpital Européen Georges Pompidou - APHP, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de St Etienne, Saint-Priest-en-Jarez
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Centre Hospitalier Universitaire Hautepierre, Strasbourg
  - Institut de Cancérologie de Lorraine - Alexis Vautrin, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No